CLINICAL TRIAL: NCT00014547
Title: Phase II Study Of BBR 3464 As Treatment In Patients With Sensitive Or Refractory Small Cell Lung Cancer After One Prior Chemotherapy Regimen
Brief Title: BBR 3464 in Treating Patients With Metastatic Small Cell Lung Cancer That Has Not Responded to Previous Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Theradex (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068555; THERADEX-TPT-II-04; NOVUSPHARMA-TPT-II-04; NCI-V01-1653
Record Dates: First submitted 2001-04-10; First posted 2004-03-11 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2002-01

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — BBR 3464

INTERVENTIONS:
Drug: BBR 3464

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BBR 3464 in treating patients who have metastatic small cell lung cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of BBR 3464 in terms of response rate in patients with sensitive or refractory metastatic small cell lung cancer. II. Determine the duration of response and time to progression in patients treated with this drug. III. Determine the overall survival of patients treated with this drug. IV. Determine the incidence and severity of toxic effects of this drug in this patient population. V. Determine the pharmacokinetics of this drug in this patient population.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (refractory vs sensitive). Patients receive BBR 3464 IV over 1 hour on day 1. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response or stable disease may receive up to 6 courses of therapy. Patients without progressive disease after 6 courses may continue treatment at the investigator's discretion. Patients are followed every 9 weeks for 3 years.

PROJECTED ACCRUAL: A total of 24-74 patients (12-37 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic small cell lung cancer (SCLC) Must have sensitive or refractory disease after first-line chemotherapy Refractory Progressive or stable disease during chemotherapy Relapse after a response during treatment Relapse after a response within 3 months after completing chemotherapy Sensitive Relapse after a response of at least 3 months duration after completing chemotherapy At least 1 measurable lesion No previously irradiated lesions No symptomatic brain or leptomeningeal metastasis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Hemoglobin at least 9 g/dL Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN ALT or AST no greater than 2.5 times ULN Albumin at least 2.5 g/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 40 mL/min (60 mL/min if treated with prior cisplatin therapy) Cardiovascular: No congestive heart failure or angina pectoris (even if medically controlled) No myocardial infarction within the past year No uncontrolled hypertension or arrhythmia Other: No other serious illness or medical condition No history of significant neurologic disorder (other than metastatic disease or psychiatric disorder) No uncontrolled infection No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer, carcinoma in situ or the cervix, or other surgically cured cancer No other condition that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy for SCLC and recovered No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for carboplatin at doses of at least 500 mg/m2 or AUC more than 7 mg/mL) and recovered No more than 1 prior chemotherapy regimen No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy for SCLC and recovered No concurrent steroids for brain metastasis No concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy except palliative local radiotherapy for non-target lesions Surgery: At least 4 weeks since prior major surgery and recovered Other: At least 30 days since prior investigational drugs and recovered No other concurrent anti-cancer therapy No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Socinski, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (18):
- United States (18):
  - Clinical Research Consultants, Inc, Hoover, Alabama
  - Highlands Oncology Group, P.A., Fayetteville, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Office of Peter D. Byeff, Southington, Connecticut
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Indiana Cancer Pavilion, Indianapolis, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - University Hospital Lexington, Lexington, Kentucky
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Theradex, Princeton, New Jersey
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Cancer Services, Columbus, Ohio
  - Oklahoma Oncology Inc., Tulsa, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Massey Cancer Center, Richmond, Virginia